CLINICAL TRIAL: NCT06630234
Title: A Master Protocol for the Multi-cohort, Open-label, Phase 1/2 Study of DCC-3009 in Participants With Gastrointestinal Stromal Tumor (GIST)
Brief Title: A Master Protocol to Evaluate DCC-3009 in Gastrointestinal Stromal Tumor (GIST)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCC-3009-01-001
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: PDGFRA mutations; KIT mutations
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DCC-3009 Module A (Experimental): Participants will receive DCC-3009 in 28 day cycles in Module A Part 1 dose escalation and Part 2 dose expansion.
  Interventions: Drug: DCC-3009

INTERVENTIONS:
Drug: DCC-3009 — Administered orally

SUMMARY:
The purpose of this Phase 1/2 master protocol study is to evaluate if DCC-3009 is safe, tolerable and works effectively in the treatment of GIST. The study will use a modular approach with each module being defined according to therapy: DCC-3009 alone or DCC-3009 in combination with other anticancer therapies. Each module will be conducted in 2 parts: Part 1 (Dose Escalation) and Part 2 (Dose Expansion). Participants will be treated in 28-day treatment cycles with an estimated duration of up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

Module A Part 1 (Escalation):

* Any participant with histologically or cytologically confirmed advanced/unresectable or metastatic GIST with documented KIT or platelet-derived growth factor receptor alpha (PDGFRA) mutation, who has progressed on or was intolerant to at least 1 approved tyrosine kinase inhibitor (TKI) regimen in the advanced/metastatic setting
* Have at least 1 measurable lesion as defined by mRECIST, v1.1
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* Adequate organ function, bone marrow function, and electrolytes
* All participants agree to comply with the contraception requirements
* Have a life expectancy of more than 3 months

Exclusion Criteria:

* Received systemic anticancer therapy or radiotherapy within 14 days prior to first dose of study drug
* Prior or concurrent malignancy that requires treatment or is expected to require treatment for active cancer
* Has known active central nervous system (CNS) metastases or an active primary CNS cancer
* History or presence of clinically relevant cardiovascular abnormalities
* Major surgery within 28 days of the first dose of study drug
* Had systemic arterial thrombotic or embolic events within 6 months prior to the first dose of study drug
* Had venous thrombotic events (e.g., deep vein thrombosis) or venous thrombotic embolic events (e.g., pulmonary embolism) within 1 month prior to the first dose of study drug
* Known allergy or hypersensitivity to any component of the study drug
* Malabsorption syndrome or other illness that could affect oral absorption
* Any other clinically significant comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities (DLT) (Part 1 Escalation) | Cycle 1 (28 Days)
  DLTs assessed for each dose level.
Objective Response Rate (ORR) (Part 2 Expansion) | Baseline to Progressive Disease (PD), Death due to Any Cause, or Start of New Antitumor Therapy (Estimated up to 24 months)
  ORR is the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR) based on Modified Response Evaluation Criteria in Solid Tumors (mRECIST), v1.1.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) (Part 1 Escalation) | Baseline to Progressive Disease (PD), Death due to Any Cause, or Start of New Antitumor Therapy (Estimated up to 24 months)
  ORR is the percentage of participants with confirmed complete response (CR) or confirmed partial response (PR) based on mRECIST, v1.1.
Duration of Response (DOR) | First Recorded CR or PR until PD or Death (Estimated up to 24 months)
  DOR for participants with confirmed CR or confirmed PR based on mRECIST, v1.1, defined as the time interval from the time that the measurement criteria are first met for CR or PR (whichever is first recorded) until the first date that the disease progression is objectively documented or death, whichever occurs first.
Progression-Free Survival (PFS) | Initiation of Treatment to PD or Death (Estimated up to 24 months)
  PFS is the time from initiation of treatment until documented disease progression per mRECIST, v1.1, or death, whichever occurs first.
Overall Survival (OS) | Initiation of Treatment to Death from Any Cause (Estimated up to 24 months)
  OS is the time from initiation of treatment to the date of death from any cause.
Pharmacokinetics (PK): Maximum observed plasma drug concentration (Cmax) | Estimated up to 24 months
  Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (10):
- United States (10):
  - HonorHealth, Scottsdate, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Vanderbilt University-Ingram Cancer Center, Nashville, Tennessee